CLINICAL TRIAL: NCT03538249
Title: Functional Characterization of Respiratory Muscles and Effects of Rehabilitation in Patients With Stable Chronic Heart Failure
Brief Title: Effects of Rehabilitation in Patients With Stable Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Zahra SADEK, Head of Physical Therapy Center, Lebanese University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0H6BKP01G84
Record Dates: First submitted 2018-04-20; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure; Aerobic Exercise; Quality of Life; Respiratory Muscle Training; Strength Training; Exercise Intolerance; Cardiac Rehabilitation
Keywords: Heart Failure; Aerobic Exercise; Respiratory Muscle Training; Strength Training
MeSH Terms: conditions — Heart Failure | interventions — Breathing Exercises; Resistance Training

STUDY DESIGN:
Intervention Model Description: Interventions Aerobic exercise training Patients follow an alternating aerobic training using a treadmill at an intensity of 60% of maximum heart rate, 3 mn and 3 mn working off an alternative way.To ensure progressive overload appropriate, we adjust moderate intensity aerobic exercise every two weeks with an overall 5% increase in heart rate.
  Inspiratory muscle training The inspiratory muscle training involves a high intensity endurance training to 60% of PI, max. We recalculate the individual SPImax and PImax in each training session. Patients use the driving tool inspiratory muscle.
  Resistance training The resistance should be measured on 1 RM (Repetition Maximum) for each muscle group. The exercises are performed in three sets of ten repetitions of exercises at 60% of 1RM intensity recalculated every two weeks training.
Who Masked: Participant, Outcomes Assessor
Masking Description: All evaluations were performed by investigators who were unaware of the allocation of patients to different interventions.

ARMS (6):
- Aerobic training (Experimental): Patients follow an alternating aerobic training using a treadmill at an intensity of 60% of maximum heart rate, 3 mn and 3 mn working off an alternative way.To ensure progressive overload appropriate, we adjust moderate intensity aerobic exercise every two weeks with an overall 5% increase in heart rate.
  Interventions: Other: Aerobic training
- Inspiratory muscle training (Experimental): The inspiratory muscle training involves a high intensity endurance training to 60% of PI, max. We recalculate the individual SPImax and PImax in each training session. Patients use the driving tool inspiratory muscle.
  Interventions: Other: Inspiratory muscle training
- Resistance training (Experimental): The resistance should be measured on 1 RM (Repetition Maximum) for each muscle group. The exercises are performed in three sets of ten repetitions of exercises at 60% of 1RM intensity recalculated every two weeks training.
  Interventions: Other: Resistance Training
- Control (No Intervention): The control group patients were allocated to a non-training time period, during which they were told to continue their life as before enrollment.
- Aerobic and Inspiratory training (Experimental): Note that the Aerobic and Inspiratory group participant undergone same protocols of inspiratory and aerobic training stated above, with almost a 5 minutes rest in between.
  Interventions: Other: Aerobic and Inspiratory training
- Combined (Experimental): Note that the Aerobic, Inspiratory and resistance group participant undergone same protocols of inspiratory and aerobic training stated above, with almost a 5 minutes rest in between.
  Interventions: Other: Combined

INTERVENTIONS:
Other: Aerobic training
  Arms: Aerobic training
Other: Inspiratory muscle training
  Other Names: Respiratory Training
  Arms: Inspiratory muscle training
Other: Resistance Training
  Other Names: Strength training
  Arms: Resistance training
Other: Aerobic and Inspiratory training
  Arms: Aerobic and Inspiratory training
Other: Combined — Aerobic, inspiratory and resistance training
  Arms: Combined

SUMMARY:
Heart failure (HF) is a major public health problem. This is the first cause of hospitalization and mortality of about 65 years old. This syndrome is characterized by a poor prognosis and a high cost of care. Thus, new strategies for treatment and prevention of the HF are among the major challenges facing health sciences today.

The management of HF requires multimodal approach it involves a combination of non-pharmacological and pharmacological treatment, Besides improvements in pharmacological treatment, supervised exercise programs are recommended for all patients with HF as part of a non-pharmacological management but many questions regarding exercise training in HF patients remain unanswered. Even simple questions such as the best mode of training for these patients are unclear.

The aim of this study

1. First, to characterize the physiological functions involved in the genesis of exercise intolerance and dyspnea especially muscle function (respiratory and skeletal), and cardiopulmonary patients suffering from chronic HF.
2. Second, to study and compare the effects of different rehabilitation programs and prove the superiority of the combination of three training modalities program: aerobic training (AT), resistance training (RT) and inspiratory muscle training (IMT).

These modalities are:

Aerobic Training: It has been proven effective in improving muscle abnormalities on changing the ventricular remodeling, dyspnea, functional capacity, increasing the maximum performance and reducing hospitalization in subjects suffering HF.

Resistance Training: It has been proven effective in improving skeletal muscle metabolism and angiogenesis; increasing capillary density and blood flow to the active skeletal muscles, promoting the synthesis and release of nitric oxide, and decreasing oxidative stress.

Selective Inspiratory Muscle Training: It has been proven effective in improving the strength and endurance of the respiratory muscles and reduction of dyspnea during daily activities.

DETAILED DESCRIPTION:
The Heart failure is the major cause of mortality and morbidity especially in elderly subjects.

The main feature of heart failure is exercise intolerance, which is always associated with fatigue and dyspnea in exercises of low intensity. Harrigton et al in 1997 demonstrated the existence of a dysfunction of skeletal muscles. But it is likely that these changes are not limited to the musculature of the lower limbs but are widespread and may affected the respiratory muscles. Thus, this dysfunction of the respiratory and skeletal muscles associated with dyspnea can contribute to the genesis of fatigue and impaired physical performance in turn reducing the autonomy of individuals.

The guidelines recommend no pharmacologic strategies by specific exercises to relieve symptoms, improve exercise tolerance and quality of life and reduce the rate of hospitalization.

The supervised exercise programs are recommended for all patients who have CHF as part of a non-pharmacological management. Thus, the exercise remains the pioneer of cardiac rehabilitation programs. The effectiveness of the training of the skeletal muscles against resistance (RT) and aerobic training (AT) in the rehabilitation HF has been well documented. However, selective training of respiratory muscles (IMT) is a relatively new technique in the field of the ICC.

In 1995, Mancini et al. were the first to publish a report on the advantage of selective training of respiratory muscles in HF patients.

Another study showed the superiority of a high-intensity training, 60% of maximal inspiratory pressure (PI max) on another 15% of PImax by increasing muscle strength and inspiratory muscle endurance, improved exercise capacity, reduction of dyspnea and quality of life.

While the above studies have investigated the benefits of inspiratory muscle training alone in CF patients, the question to ask is "If the benefit of the inspiratory muscle training was added to that observed with aerobic training for the whole body. "

Laoutaris in 2013 showed that the combination of AT with RT and IMT could result in a significant improvement in peripheral muscle and respiratory function with significant improvement in exercise capacity, dyspnea and quality of life compared to that of the 'single AT. However, this study has several limitations. These limits are:

1. Patients in the combined group suffer longer exercise sessions of 20 minutes compared to patients alone aerobic group. Thus, the difference in the time to exercise between the 2 groups may have influenced the results of the study.
2. Furthermore, the authors compared three different modalities of exercising against a modality which affects so the quality of the study.
3. In addition, the extent to which the resistance training or selective training of respiratory muscles contributed to greater improvements in the combined group was not assessed in this study as this would take several modalities groups different exercises and a control group.

Till now,

1. There are no randomized, controlled, double blinding studies that compares different modalities of exercises to each other and to a control group in patients who have CHF. Moreover,
2. It is not known until now what combination of exercises modalities is the most effective and more secure, and
3. If there are additional benefits by combining multiple training modalities by comparing it with other modalities in patients with stable chronic heart failure (CHF).

In this study, the investigators examined the hypothesis of the efficiency of a combined program of three modalities: aerobics, resistance, and selective respiratory muscle on:

1. Heart and lung function,
2. Heart and lung structure,
3. The function of skeletal and respiratory muscles,
4. Functional capacity,
5. Dyspnea, and quality of life.

The main objectives of this project are defined:

1. To characterize the physiological functions involved in the genesis of exercise intolerance and dyspnea.
2. Comparative study of all therapeutic modalities with a control group and each other.
3. To study muscle function: respiratory and skeletal in HF patients in different training groups.
4. To study the muscular structures: respiratory and skeletal.
5. To study the structure and heart function.
6. See the influence of these three training modalities on functional capacity, dyspnea and quality of life.
7. To state the guidelines for heart failure.

Methodology and research requirements Protocol All subjects must sign an informed consent form. Patients will submit a physical examination, and electrocardiographic measurements by a cardiologist. Approximately 60 patients are divided randomly by investigators who are not involved in the implementation of the project to eight different groups.

Before and after the intervention were evaluated all the tests mentioned above by a physiotherapist who do not know the distribution of patients to different interventions.

Groups All types of training sessions are individualized and are carried in Beirut Cardiac Institute. Patients are exerted for twelve weeks at a rate of three times per week, for one hour. Any missed session will be added to the end of the program, so that the 36 sessions will be realized. All sessions must be supervised at all times by a physiotherapist and a cardiologist.

Group 1 (n = 10): Aerobic training (30mn) Group 2 (n = 10): Inspiratory muscle training (20mn) Group 3 (n = 10): Resistance Training (20mn) Group 4 (n = 10): Aerobic Training (30 min) + Inspiratory muscle training (20mn) Group 5 (n = 10): Aerobic Training (30 min) + Inspiratory muscle training (20minutes) + Resistance training (20 minutes) Group 6 (n = 10) Control

ELIGIBILITY:
Inclusion Criteria

* Congestive heart failure (CHF) due to ischemic or dilated cardiomyopathy.
* Left ejection fraction ≤ 45%.
* NYHA functional class II and III.
* A patient with a diagnosis of CHF for six months including no admission to the hospital or change in medications over the previous 3 months.
* IMW <70% of predicted

Exclusion criteria

* Pulmonary limitation (forced expiratory volume in 1 s and/or vital capacity of less than 60% of predicted value).
* History of significant cardiac arrhythmia.
* History of myocardial infarction or cardiac surgery (6 months).
* Orthopedic or neurologic disease.
* Non echogenic, Unstable.
* Poorly controlled blood pressure.
* End-Stage HF (on the waiting list for transplantation or LVAD).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10-15 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Minnesota Living with Heart Failure Questionnaire (MLWHF) | Baseline and 12 weeks
  The Quality of life was assessed using the Minnesota Living with Heart Failure Questionnaire (MLWHF). the minimum score is 0 and the maximum score is 105. the total score should decrease to indicate the amelioration of the quality of life.

SECONDARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | Baseline and 12 weeks
  FVC was assessed to evaluate the lung Function. FVC measurement shows the amount of air a person can forcefully and quickly exhale after taking a deep breath.
Change in Forced Expiratory Muscle Volume in one second (FEV1) | Baseline and 12 weeks
  FEV1 was assessed to evaluate the lung Function. FEV1 measurement shows the amount of air a person can forcefully exhale in one second of the FVC test.
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline and 12 weeks
  LVED was assessed to evaluate the cardiac function by using echocardiography at rest. LVEF (%) : the total amount of blood in the left ventricle is pumped out with each heartbeat.
Change in Left Ventricular End Systolic and Diastolic Diameter (LVESD and LVEDD) | Baseline and 12 weeks
  LVESD and LVEDD was assessed to evaluate the cardiac function by using echocardiography at rest. Evaluation of the Left Ventricule dimensions (mm) and wall thicknesses in end-systolic and end-diastolic.
Change in Maximal Inspiratory Pressure (MIP) | Baseline and 12 weeks
  MIP (cm h2o) was assessed to evaluate the strength of inspiratory muscles using Electronic pressure transducer.
Change in Sustained Maximal Inspiratory Pressure [SMIP] | Baseline and 12 weeks
  SMIP (Secondes) was used to assess the respiratory muscle endurance where the time was recorded in the period during which a patient can cover maintaining 70% MIP.
Change in Borg scale | Baseline and 12 weeks
  The dyspnea was assessed using Borg Scale. the minimum score is 6 and the maximum score is 20. the total score should decrease to indicate the amelioration of the dyspnea.
Change in six-minute walk test (6MWT) | Baseline and 12 weeks
  The Functional capacity was assessed by using 6MWT in meters. the distance should increase to indicate the amelioration of the functional capacity.
Change in Exercise time in stress test | Baseline and 12 weeks
  Exercise time (secondes) was assessed using Stress test on a treadmill according to the Bruce protocol. the time should increase to indicate the amelioration of the aerobic capacity.
Change in Metabolic Equivalent of a Task (METs) | Baseline and 12 weeks
  The assessment of workload is measured by METs during stress test. METs is a unit that estimates the amount of energy used by the body during physical activity, as compared to resting metabolism. The unit is standardized so it can apply to people of varying body weight and compare different activities.
Change in Maximal Voluntary Isometric Force (MVIF) | Baseline and 12 weeks
  MVIF (Kg) was assessed to evaluate the function of skeletal muscles using Dynamometer; to assess the strength of the quadriceps muscle.
Change in Isometric endurance time (MT) | Baseline and 12 weeks
  MT (secondes) was assessed to evaluate the endurance of the quadriceps muscle. MT was measured when subjects maintained an isometric contraction at 50% of the reported MVIF.

IPD SHARING:
Plan to Share IPD: Undecided
no plan

REFERENCES:
- [Derived] Sadek Z, Salami A, Youness M, Awada C, Hamade M, Joumaa WH, Ramadan W, Ahmaidi S. A randomized controlled trial of high-intensity interval training and inspiratory muscle training for chronic heart failure patients with inspiratory muscle weakness. Chronic Illn. 2022 Mar;18(1):140-154. doi: 10.1177/1742395320920700. Epub 2020 May 5. PMID 32370544